CLINICAL TRIAL: NCT02109172
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Cross-Over Study of QD and BID Nebulized TD-4208 in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 7-Day Cross-over Study of QD (Once Daily) and BID (Twice Daily) TD-4208 in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0116
Record Dates: First submitted 2014-04-06; First posted 2014-04-09 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TD-4208 44 mcg twice daily (Experimental): TD-4208 inhalation solution 44 mcg twice daily for 7 days
  Interventions: Drug: TD-4208
- Placebo (Placebo Comparator): Placebo inhalation solution twice daily for 7 days
  Interventions: Drug: Placebo
- TD-4208 175 mcg once daily (Experimental): TD-4208 inhalation solution 175 mcg once daily, placebo once daily
  Interventions: Drug: TD-4208; Drug: Placebo

INTERVENTIONS:
Drug: TD-4208
  Other Names: Revefenacin
  Arms: TD-4208 175 mcg once daily; TD-4208 44 mcg twice daily
Drug: Placebo
  Arms: Placebo; TD-4208 175 mcg once daily

SUMMARY:
This study evaluated the safety and efficacy of once and twice daily TD-4208 and placebo when administered using a jet nebulizer for 7 days in a cross-over design to patients with moderate to severe chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a negative pregnancy test, and must be prepared to use effective contraception if of child-bearing potential
* Subject is capable of performing reproducible spirometry maneuvers
* Subject has post-bronchodilator FEV1/FVC (forced expiratory volume in 1 second/forced vital capacity) ratio <0.7
* Subject has moderate-to-severe stable COPD (Stage 2 or 3 according to the Global Initiative for the Treatment of Obstructive Lung Disease (GOLD) Guidelines)
* Subject has a post-bronchodilator FEV1 greater than or equal to 30% and less than 80% of predicted normal
* Subject demonstrates a post-ipratropium FEV1 response ≥ 12% and ≥ 200 mL of pre-ipratropium FEV1 response
* Subject has a current or past smoking history of at least 10 pack-years.

Exclusion Criteria:

* Subject has a significant respiratory disease or disorder other than COPD that would affect the interpretation of data from this study
* Subject has a history of reactions or hypersensitivity to inhaled anticholinergic or beta-agonist agents
* Subject suffers from any medical condition that would preclude the use of inhaled anticholinergic agents
* Subject has been hospitalized for COPD or pneumonia within 12 weeks.
* Subject requires long-term oxygen therapy (>15 hours a day)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma, US, Inc.
Locations (1):
- American Health Research, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then 44mcg, Then 175mcg: Placebo twice daily for 7 days then 44mcg twice daily for 7 days then 175mcg once daily for 7 days
- Placebo First, Then 175mcg, Then 44mcg: Placebo twice daily for 7 days then 175mcg once daily for 7 days then 44mcg twice daily for 7 days
- 44mcg First, Then 175mcg, Then Placebo: 44mcg twice daily for 7 days then 175mcg once daily for 7 days then placebo twice daily for 7 days
- 44mcg First, Then Placebo, Then 175mcg: 44mcg twice daily for 7 days then placebo twice daily for 7 days then 175mcg once daily for 7 days
- 175mcg First, Then 44mcg, Then Placebo: 175mcg once daily for 7 days then 44mcg twice daily for 7 days then placebo twice daily for 7 days
- 175mcg First, Then Placebo, Then 44mcg: 175mcg once daily for 7 days then placebo twice daily for 7 days then 44mcg twice daily for 7 days
Period: Overall Study
Arm/Group | Placebo First, Then 44mcg, Then 175mcg | Placebo First, Then 175mcg, Then 44mcg | 44mcg First, Then 175mcg, Then Placebo | 44mcg First, Then Placebo, Then 175mcg | 175mcg First, Then 44mcg, Then Placebo | 175mcg First, Then Placebo, Then 44mcg
Started | 11 | 11 | 10 | 11 | 10 | 11
Completed | 10 | 11 | 9 | 10 | 9 | 10
Not Completed | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All groups were randomized to receive placebo, TD-4208 44mcg twice daily, and TD-4208 175 mcg once daily
Arm/Group | Entire Study Population
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean (0-24hr) Change From Baseline FEV1 (Forced Expiratory Volume in 1 Second)
Description: Weighted mean (0-24hr) Change from baseline FEV1 (forced expiratory volume in 1 second). Measurement is change from baseline.
Time Frame: Following the Day 7 AM dose -12 hours post-dose and 24 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: mL
Groups:
- Placebo: Placebo inhalation solution twice daily for 7 days
  Placebo
- TD-4208 44 mcg Twice Daily: TD-4208 inhalation solution 44 mcg twice daily for 7 days
  TD-4208
- TD-4208 175 mcg Once Daily: TD-4208 inhalation solution 175 mcg once daily, placebo once daily
  TD-4208
  Placebo
Arm/Group | Placebo | TD-4208 44 mcg Twice Daily | TD-4208 175 mcg Once Daily
Number analyzed (Participants) | 64 | 64 | 64
mL | -14.4 (15.29) | 90.2 (15.00) | 98.5 (15.03)

ADVERSE EVENTS:
Groups:
- TD-4208 44mcg Twice Daily: TD-4208 inhalation solution 44 mcg twice daily for 7 days
- TD-4208 175mcg Once Daily: TD-4208 inhalation solution 175 mcg once daily
Arm/Group | Placebo | TD-4208 44mcg Twice Daily | TD-4208 175mcg Once Daily
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 1/64
Other Adverse Events (participants affected / at risk) | 23/64 | 24/64 | 14/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | TD-4208 44mcg Twice Daily (N=64) | TD-4208 175mcg Once Daily (N=64)
Coronary Artery Insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | TD-4208 44mcg Twice Daily (N=64) | TD-4208 175mcg Once Daily (N=64)
Blood Pressure Increased (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Coronary artery insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was designed to evaluate whether a lower dose (44) BID would achieve a greater response than a higher dose (175) QD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.